CLINICAL TRIAL: NCT00567632
Title: Generation of Standard Laboratory Values for Pneumococci Antibodies
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Markus A. Rose, ass. Professor of Paediatrics, Goethe University, Childrens' Hospital
Other Study IDs: 1-Rose
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2007-10

CONDITIONS: Reference Values
Keywords: Pneumococci; Antibody; Standard laboratory values

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The determination of reference values is a necessary basis for research and clinical routine testing for pneumococci antibodies

DETAILED DESCRIPTION:
This study is meant to determine specific pneumococcal antibodies stratified for age. The investigators also correlate our assay with the results from a commercially available pneumococcal screening ELISA (iGG1 and IgG2) in order to facilitate a screening for immunodeficiency, and to monitor the success of a performed immunization

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing elective surgery

Exclusion Criteria:

* Chronic illness condition,
* Immunodeficiency

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: any clinically and immunologically healthy subject of any age undergoing selective surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
sufficient samples to calculate reference values | 10(2006-10/2007)

SECONDARY OUTCOMES:
sufficient samples to correlate with screening assay | 10/2006-10/2007

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Rose, M.D., Ph.D., M.P.H, Study Chair — Goethe University, childrens Hospital
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany